CLINICAL TRIAL: NCT04101734
Title: Thyromental Height Test as a New Method for Prediction of Difficult Intubation Using Double Lumen Video Tubes
Brief Title: TMHT - Difficult Intubation Prediction Using Double Lumen Video Tubes
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: TMHT-04
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Predictive Value of Tests; Intubation;Difficult
Keywords: Difficult Intubation; Thyromental Height Test; Double Lumen Video Tube

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Double Lumen Endotracheal Tube: Group of patients intubated with Double Lumen Endotracheal Tube.
  Interventions: Device: Double Lumen Endotracheal Tube.
- Double Lumen Video Endotracheal Tube: Group of patients intubated with Double Lumen Video Endotracheal Tube.
  Interventions: Device: Double Lumen Video Endotracheal Tube.

INTERVENTIONS:
Device: Double Lumen Endotracheal Tube. — Intubation was performed with Double Lumen Endotracheal Tube.
  Groups: Double Lumen Endotracheal Tube
Device: Double Lumen Video Endotracheal Tube. — Intubation was performed with Double Lumen Video Endotracheal Tube.
  Groups: Double Lumen Video Endotracheal Tube

SUMMARY:
The purpose of this study is to assess the usefulness of the Thyromental Height Test in prediction of difficult intubation and the utility of double lumen video endotracheal tubes in patients scheduled for elective thoracic procedures.

DETAILED DESCRIPTION:
Most of the thoracic surgery interventions require lung isolation techniques. Currently the most commonly used lung isolation techniques are double lumen tubes or single lumen tubes with additional use of bronchial blockers. In both cases fiberoptic bronchoscopy is used for proper placement and maintenance during operation. Recently double lumen video endotracheal tubes were proposed as a new alternative for lung isolation techniques. The double lumen video endotracheal tube differs significantly in size and physical characteristics from standard single lumen endotracheal tube and intubation may prove to be challenging even for an experienced practitioner. Therefore proper prediction of difficult intubation play a crucial role in a clinical setting. Sensitivity and specificity of existing anthropometric scales and tests used for prediction of difficult intubation seem lacking so new methods such as Thyromental Height Test (TMHT) are being introduced. It is based on the height between the anterior border of the thyroid cartilage and the anterior border of the mentum, measured while the patient lies in the supine position with closed mouth. The main objective of the trial is to assess the clinical usefulness of TMHT in prediction of difficult intubation using double lumen video endotracheal tubes in patients scheduled for elective thoracic surgical procedures. The secondary aim is to evaluate the utility of double lumen video endotracheal tubes as a novel method of lung separation.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective thoracic procedures, requiring general anaesthesia and intubation with double lumen endotracheal tubes
* written, informed consent for participation in the trail
* older than 18 years

Exclusion Criteria:

* emergency procedures
* visible anatomic abnormalities
* patients scheduled for awake fibre optic intubation
* lack of consent for participation in the trail

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing elective thoracic procedures in university hospital, requiring general anaesthesia and intubation with a double lumen endotracheal tubes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Thyromental height | Preoperative (1 day prior to the operation)
  The height between the anterior border of the thyroid cartilage (on the thyroid notch just between the 2 thyroid laminae) and the anterior border of the mentum (on the mental protuberance of the mandible), in supine position with mouth closed, measured with a depth gauge during routine preoperative anaesthetic visit.

SECONDARY OUTCOMES:
Time of Intubation | Intraoperatively
  Time of intubation defined as a time from direct laryngoscopy to proper placement of double lumen endotracheal tube measured with a timer during induction of general anesthesia.
Airway trauma | Intraoperative
  During fiberoptic bronchoscopy after the operation airway trauma on the level of bronchus, tracheal bifurcation, trachea and vocal cords were reported, where 0 was defined as no visible trauma, 1 as a redness, 2 as oedema, 3 as hematoma and 4 as active bleeding.
Usage of fiberoptic bronchoscopy | Intraoperatively
  Usage of fiberoptic bronchoscopy for proper placement of double lumen tube was noted.
score in Cormack-Lehane scale | Preoperative (1 day prior to the operation)
  During direct laryngoscopy the laryngeal view is graded in Cormack-Lehane Scale by the laryngoscopist. Grade I is assigned when the glottis is fully visible, grade II when the glottis is partially visible, grade III when only the epiglottis is visible and grade IV when neither glottis nor epiglottis is visible.
Thyromental distance | Preoperative (1 day prior to the operation)
  The distance between the thyroid prominence and the most anterior part of the mental prominence of the mandible, measured with a standard centigrade ruler as the distance in centimetres with the patient in supine position, head fully extended, mouth closed, during routine preoperative anaesthetic visit.
Sternomental distance | Preoperative (1 day prior to the operation)
  The distance in centimetres between the superior border of the manubrium sterni and the bony point of the mentum, with the patient in supine position, head fully extended, mouth closed, measured with a standard centigrade ruler, during routine preoperative anaesthetic visit.
score in modified Mallampati test | Preoperative (1 day prior to the operation)
  The oropharyngeal view is assessed in sitting position, mouth maximally opened, tongue protruded, without phonation, measured during routine preoperative anaesthetic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Misiołek, MD PhD, Study Director — Medical University of Silesia; Szymon Białka, MD, Study Chair — Medical University of Silesia
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland

REFERENCES:
- [Derived] Palaczynski P, Misiolek H, Bialka S, Owczarek AJ, Gola W, Szarpak L, Smereka J. A randomized comparison between the VivaSight double-lumen tube and standard double-lumen tube intubation in thoracic surgery patients. J Thorac Dis. 2022 Oct;14(10):3903-3914. doi: 10.21037/jtd-22-451. PMID 36389329